CLINICAL TRIAL: NCT05309642
Title: Effect of 12-week Intermittent Calorie Restriction on Liver Fat Content in Comparison With Standard-of-care in Patients With Nonalcoholic Fatty Liver Disease: a Randomized Controlled Trial
Brief Title: Nonalcoholic Fatty Liver Disease - Intermittent Calorie Restriction (FLICR) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Hwi Young Kim, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLICR
Record Dates: First submitted 2022-03-12; First posted 2022-04-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; MRI-PDFF; MR-Elastography; Intermittent Calorie Restriction; Liver metabolite; Gut microbiome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomly allocated two groups; ICR (intermittent calorie restriction) group and SoC (standard-of-care) group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICR Arm (Active Comparator): On 2 non-consecutive days per week, participants in the ICR (5:2 diet) group will be instructed to consume 500 kcal/day for women and 600 kcal/day for men.
  Interventions: Behavioral: Intermittent calorie restriction
- Soc Arm (Placebo Comparator): The SoC group will receive 80% of standard calorie (1,200-1,500 kcal/day or reducing 500-1000 kcal/day from standard calorie).
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Intermittent calorie restriction — Recipes will be provided with suggestions of meals that would not exceed the calorie restriction. For the remaining 5 days of the week, they will receive instructions and recipes that follows the Korean Dietary Reference Intakes (KDRIs), with an intake limit of 2,000 kcal/day for women and 2,500 kcal/day for men. The percentage of energy (E%) from different macronutrients in the recipes will be 45-60 E% carbohydrates, 25 E% fat and 10-20 E% protein.
  Arms: ICR Arm
Behavioral: Standard of care — They will receive individualized guidance from a hepatologist on how to choose a healthy diet, to reduce the intake of sweets and saturated fatty acids, increase sources of unsaturated fat, avoid large portions, and to regularly eat 3 meals per day. Each participant will be provided a written summary of the dietary advice.
  Arms: Soc Arm

SUMMARY:
Several diets have been proposed to reduce liver steatosis in patients with nonalcoholic fatty liver disease (NAFLD), and various effects on liver steatosis have been observed. The objective of this trial is to compare the effects of intermittent calorie restriction (ICR) (5:2 diet) and standard-of-care (SoC) on reduction of hepatic steatosis.

DETAILED DESCRIPTION:
This is an open-label randomised controlled trial of patients with NAFLD. Patients are recruited in the Liver Outpatient Clinic of the Ewha Womans University Mokdong Hospital. The department of Nutritional Science and Food Management, Ewha Womans University will collaborate for this study.

About 72 patients (36 patients with body mass index [BMI] ≥25 kg/m2 and 36 patients with BMI <25 kg/m2) will be enrolled in a 1:1 ratio to 12 weeks treatment with either 5:2 diet (ICR group, 18 patients in each BMI group), or general lifestyle advice from a hepatologist (standard of care; SoC group, 18 patients in each BMI group).

Beginning in week 3 (Visit 2), an ICR group and a SoC group are generated through randomisation. Both arms will be accompanied for a duration of 12 weeks. After 12 weeks from the completion of the experimental phase (wash-out period), there will be the "end of follow up" visit.

The whole duration of the study is 26 weeks (2 weeks lead-in, 12 weeks intervention and 12 weeks post-intervention investigation).

Magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) and MR-Elastography are conducted at the screening visit and at weeks 12.

There will be 5 visits at the study center (screening, randomization, week 8, end of treatment and end of study) and 10 phone visits (week 4, 5, 6, 7, 8, 10, 11, 12, 13, 14). At each visit clinical events, anthropometric index and standard laboratory parameters will be collected. Participants will fill in questionnaires capturing quality of life.

Adverse events will be recorded. Phone visits are used to survey the safety of patients.

Non-adherence to ICR for 20% of the total study period has been selected as cut off to define treatment failure at per-protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

1. NAFLD diagnosed by (1) Histologic assessment with a fat accumulation of more than 5% of the liver's weight in a biopsy, or (2) Radiologic assessment with a MRI-PDFF ≥8%.
2. Age between 19 and 75 years
3. Capability to understand the study and the individual consequences of participation
4. Signed and dated declaration of agreement in the forefront of the study

Exclusion Criteria:

1. Daily alcohol consumption >30 g in men and >20 g in women
2. Other causes of chronic liver disease (HBV, HCV, HDV, HEV, HIV), autoimmune diseases or chronic cholestatic liver disease, drug induced liver injury, hereditary haemochromatosis, Wilson disease, α-1-Antitrypsin deficiency
3. Liver cirrhosis
4. Hepatocellular carcinoma
5. Medications which cause liver disease or secondary NAFLD (e.g. Tamoxifen, systemic Corticosteroids, Methotrexate, Tetracycline, Estrogens, Valproic acid)
6. Changes in body weight > 5% in the last 3 months
7. Intake of medical treatment for NAFLD/NASH in the last 6 months (except for vitamin E)
8. Diabetes
9. Pregnancy
10. Patients after organ transplantations
11. Missing or lacking consent capability

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Impact of ICR on liver steatosis by MRI-PDFF | Baseline, 12 weeks
  The primary outcome of interest is a change in MRI-PDFF value of a least 30% with ICR

SECONDARY OUTCOMES:
Changes in liver fibrosis by MR-Elastography | Baseline, 12 weeks
  Measure the change of liver fibrosis with MR-Elastography
Changes in anthropometrics | Baseline, 12, and 24 weeks
  BMI (kg/m2)
Changes in body composition analysis (BCA) | Baseline, 12, and 24 weeks
  Measure the change of BCA with Inbody
Changes in visceral adipose tissue (VAT) | Baseline, 12, and 24 weeks
  Measure the change of VAT with fat CT
Changes in quality of life score | Baseline, 12, and 24 weeks
  Measure the change of Quality of Life score with Chronic Liver Disease-NAFLD questionnaire (CLDQ). The CLDQ uses 29 items in four domains, each scored on a Likert scale from 1 (all of the time) to 7 (none of the time) representing the frequency of clinical symptoms and emotional problems in the last two weeks. Results are reported in the six subscale scores (abdominal symptoms, fatigue, systemic symptoms, activity, emotional functioning, worry) and a CLDQ overall score.
Genetic analysis | Baseline
  Polymorphism of PNPLA3, TM6SF2, TM4SF5, SREBF2, MBOAT7-TMC4, HSD17B13 and adenine insertion (A-INS) will be analyzed by NGS (Next Generation Sequencing)
Changes in hormone | Baseline, 12 weeks
  Measure the change of leptin, adiponectin, ghrelin, GLP-1, apelin, and osteopontin
Changes in liver metabolite | Baseline, 12 weeks
  Measure the change of diglycerides (DG), FA, phosphatidylethanolamines (PE), phosphatidylcholines (PC), methionine, SAMe, and methylthioadenosine
Changes in gut microbiota | Baseline, 12 weeks
  Evaluation of 16S rRNA gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Hwi Young Kim, Professor, Principal Investigator — Ewha Womans University College of Medicine
Locations (1):
- Ewha Womans University College of Medicine, Seoul, Yangcheon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmer M, Lindqvist C, Petersson S, Moshtaghi-Svensson J, Tillander V, Brismar TB, Hagstrom H, Stal P. Treatment of NAFLD with intermittent calorie restriction or low-carb high-fat diet - a randomised controlled trial. JHEP Rep. 2021 Feb 17;3(3):100256. doi: 10.1016/j.jhepr.2021.100256. eCollection 2021 Jun. PMID 33898960
- [Background] Younossi ZM, Corey KE, Lim JK. AGA Clinical Practice Update on Lifestyle Modification Using Diet and Exercise to Achieve Weight Loss in the Management of Nonalcoholic Fatty Liver Disease: Expert Review. Gastroenterology. 2021 Feb;160(3):912-918. doi: 10.1053/j.gastro.2020.11.051. Epub 2020 Dec 9. PMID 33307021
- [Background] Schubel R, Nattenmuller J, Sookthai D, Nonnenmacher T, Graf ME, Riedl L, Schlett CL, von Stackelberg O, Johnson T, Nabers D, Kirsten R, Kratz M, Kauczor HU, Ulrich CM, Kaaks R, Kuhn T. Effects of intermittent and continuous calorie restriction on body weight and metabolism over 50 wk: a randomized controlled trial. Am J Clin Nutr. 2018 Nov 1;108(5):933-945. doi: 10.1093/ajcn/nqy196. PMID 30475957
- [Background] Retterstol K, Svendsen M, Narverud I, Holven KB. Effect of low carbohydrate high fat diet on LDL cholesterol and gene expression in normal-weight, young adults: A randomized controlled study. Atherosclerosis. 2018 Dec;279:52-61. doi: 10.1016/j.atherosclerosis.2018.10.013. Epub 2018 Oct 17. PMID 30408717
- [Background] Wong VW, Wong GL, Chan RS, Shu SS, Cheung BH, Li LS, Chim AM, Chan CK, Leung JK, Chu WC, Woo J, Chan HL. Beneficial effects of lifestyle intervention in non-obese patients with non-alcoholic fatty liver disease. J Hepatol. 2018 Dec;69(6):1349-1356. doi: 10.1016/j.jhep.2018.08.011. Epub 2018 Aug 22. PMID 30142427
- [Background] Cai H, Qin YL, Shi ZY, Chen JH, Zeng MJ, Zhou W, Chen RQ, Chen ZY. Effects of alternate-day fasting on body weight and dyslipidaemia in patients with non-alcoholic fatty liver disease: a randomised controlled trial. BMC Gastroenterol. 2019 Dec 18;19(1):219. doi: 10.1186/s12876-019-1132-8. PMID 31852444
- [Background] Klempel MC, Kroeger CM, Bhutani S, Trepanowski JF, Varady KA. Intermittent fasting combined with calorie restriction is effective for weight loss and cardio-protection in obese women. Nutr J. 2012 Nov 21;11:98. doi: 10.1186/1475-2891-11-98. PMID 23171320
- [Background] Carter S, Clifton PM, Keogh JB. Effect of Intermittent Compared With Continuous Energy Restricted Diet on Glycemic Control in Patients With Type 2 Diabetes: A Randomized Noninferiority Trial. JAMA Netw Open. 2018 Jul 6;1(3):e180756. doi: 10.1001/jamanetworkopen.2018.0756. PMID 30646030
- [Derived] Lee HA, Moon H, Kim Y, Lee JK, Lee HA, Kim HY. Effects of Intermittent Calorie Restriction in Nondiabetic Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease. Clin Gastroenterol Hepatol. 2025 Jan;23(1):114-123.e13. doi: 10.1016/j.cgh.2024.06.051. Epub 2024 Aug 23. PMID 39181426
- [Derived] Lee HA, Moon H, Kim Y, Lee HA, Kim HY. Effect of 12-week intermittent calorie restriction compared to standard of care in patients with nonalcoholic fatty liver disease: a randomized controlled trial. Trials. 2023 Aug 2;24(1):490. doi: 10.1186/s13063-023-07444-4. PMID 37533096